CLINICAL TRIAL: NCT06776978
Title: La Stimolazione Transcranica (tDCS) E Transpinale a Corrente Diretta (tsDCS) Per Il Recupero Delle Funzioni Cognitive in Soggetti Affetti Da Patologia Cerebrovascolare O Neurodegenerativa
Brief Title: Effectiveness of TDCS Over Broca's Area in Verb Naming: a Randomized, Double-Blind, Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CE/prog.733
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Aphasia Non Fluent; Stroke
Keywords: Transcranial Direct Current Stimulation; Aphasia; Verb Naming; Language Rehabilitation; Speech Therapy; Stroke
MeSH Terms: conditions — Aphasia, Broca; Stroke; Aphasia; Communication Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Experimental): Participants receive anodic tDCS over Broca's area at 2 mA for 20 minutes per session, 5 days per week for 2 consecutive weeks.
  Interventions: Device: Active treatment
- Sham tDCS (Sham Comparator): Participants receive sham tDCS for 20 minutes per session, 5 days per week for 2 consecutive weeks.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Active treatment — Participants receive anodic tDCS using a battery-driven Eldith (neuroConn GmbH) Programmable Direct Current Stimulator with surface-soaked sponge electrodes (5×7 cm). A constant current of 2 mA is applied for 20 minutes per session. The stimulation targets the left frontal region (F5 of the extended International 10-20 EEG system), corresponding to Broca's area, while the reference electrode is placed over the contralateral frontopolar cortex. tDCS is performed for 10 daily sessions over two consecutive weeks (5 days per week).
  Arms: Active tDCS
Device: Sham Stimulation — Participants receive sham tDCS using a battery-driven Eldith (neuroConn GmbH) Programmable Direct Current Stimulator with surface-soaked sponge electrodes (5×7 cm). No therapeutic current is applied during the 20-minute session. The electrode placement mimics the active condition, targeting the left frontal region (F5 of the extended International 10-20 EEG system), corresponding to Broca's area, while the reference electrode is placed over the contralateral frontopolar cortex. Sham tDCS is performed for 10 daily sessions over two consecutive weeks (5 days per week).
  Arms: Sham tDCS

SUMMARY:
This clinical trial investigated whether transcranial direct current stimulation (tDCS) over Broca's area (F5) could improve verb naming abilities in adults with aphasia. Additionally, the study evaluated the stability of the treatment response to tDCS over time.

The main questions this study sought to answer were:

* Does tDCS improve verb naming abilities compared to inactive (sham) stimulation?
* Are the observed effects stable over time?

Participants received 10 daily sessions of tDCS over two consecutive weeks (5 days per week). The study included two treatment conditions, separated by one-month washout period:

* Active tDCS: Stimulation over Broca's area at 2 mA;
* Sham tDCS: Stimulation mimicking the active condition without delivering electrical current.

During the treatment, participants were asked to name aloud videos of actions displayed on a computer screen. One month after each treatment condition, follow-up testing was conducted to evaluate the stability of the treatment response.

ELIGIBILITY:
Inclusion Criteria:

* native Italian proficiency;
* pre-morbid right-handedness;
* a single left hemispheric stroke at least 6 months before the investigation.

Exclusion Criteria:

* acute or chronic neurological symptoms requiring medication;
* attention and/or memory deficits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Action Naming Task | Verb naming performance was assessed at baseline (pre-treatment), post-treatment (immediately after the 10-day intervention), and at follow-up (one month after each treatment condition) to evaluate both immediate effects and the stability of responses.
  An action naming task was designed to evaluate verb naming performance. Video clips depicting various actions were presented on a 15-inch computer screen at a viewing distance of 1 meter, each preceded by an 800-millisecond fixation point. Participants were instructed to name the action depicted in each clip within a 15-second response window. The examiner manually recorded correct responses. For incorrect responses or failures to respond within the allotted time, the written name of the action was displayed beneath the video, and participants were required to read the name aloud. The video and the written name remained on the screen until the word was read correctly or 40 seconds had elapsed. The task was conducted during 20-minute tDCS sessions, wherein participants received either active stimulation targeting Broca's area or sham stimulation with identical electrode placement but no active current.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Caltagirone, MD, PhD, Principal Investigator — Fondazione Santa Lucia, Via Ardeatina 306, 00179 Roma, Italy
Locations (1):
- I.R.C.C.S. Fondazione Santa Lucia, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Syka J, Melichar I. The effect of loop diuretics upon summating potentials in the guinea pig. Hear Res. 1985;20(3):267-73. doi: 10.1016/0378-5955(85)90031-0. PMID 3003019
- [Background] Nishitani N, Schurmann M, Amunts K, Hari R. Broca's region: from action to language. Physiology (Bethesda). 2005 Feb;20:60-9. doi: 10.1152/physiol.00043.2004. PMID 15653841
- [Background] Marangolo P, Fiori V, Di Paola M, Cipollari S, Razzano C, Oliveri M, Caltagirone C. Differential involvement of the left frontal and temporal regions in verb naming: a tDCS treatment study. Restor Neurol Neurosci. 2013;31(1):63-72. doi: 10.3233/RNN-120268. PMID 23142815